CLINICAL TRIAL: NCT02425514
Title: Evaluation of Bone Union Following Anterior Cervical Fusion Using a Bioactive Glass-Ceramic Spacer (NovoMax™): Comparison With a PEEK Cage Filled With β-Tricalcium Phosphate (Cervios ChronOs™)
Brief Title: Evaluation of Bone Union Following Anterior Cervical Fusion Using a NovoMax™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioAlpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA04-CP11
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Intervertebral Disk Degeneration; Intervertebral Disk Displacement
Keywords: Anterior cervical discectomy and fusion; NovoMax; Bioactive Glass-ceramic Intervertebral Spacer
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Treatment group: Bioactive Glass-Ceramic Spacer (NovoMax™) Active comparator: a PEEK cage Filled with β-Tricalcium Phosphate
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervios ChronOs (Experimental): The ACDF surgery will be carried out with Cervios ChronOs(TM), which is the PEEK cage filled with b-TCP.
  Interventions: Device: Cervios ChronOs
- NovoMax™ (Experimental): The ACDF surgery will be carried out with NovoMax™, which is the bioactive glass ceramic intervertebral spacer
  Interventions: Device: NovoMax™

INTERVENTIONS:
Device: Cervios ChronOs — The ACDF surgery will be carried out with Cervios ChronOs after randomization procedure.
  Arms: Cervios ChronOs
Device: NovoMax™ — The ACDF surgery will be carried out with NovoMax™ after randomization procedure.
  Arms: NovoMax™

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of NovoMax™ in Anterior Cervical Interbody Fusion - Comparison of NovoMax™ versus ChronOs®.

ELIGIBILITY:
Inclusion Criteria:

* The patient who is expected to receive anterior cervical discectomy and fusion operation.
* Volunteer for this study with written consent.

Exclusion Criteria:

* Patient with cervical spine fracture, infection and malignant tumor
* Below -3.5 T-score by DEXA bone densitometry
* Patient who is not suitable for this study judged by principal investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Bone Fusion With CT and Dynamic radiographs(X-ray)(Post operative 6 Months) | at 6 months after surgery (ACDF)
  Evaluation of bone fusion between bone substitutes and cervical vertebral endplates with 3-dimensional CT and X-ray at 6 months after operation (ACDF).

SECONDARY OUTCOMES:
VAS of Neck Pain(Post operative 6 Months) | at 6 months after surgery (ACDF)
  Evaluation of neck pain using the visual analogue scale (VAS) at 6 months after operation (ACDF). Reported pain using VAS was recorded and evaluated. Patients were instructed to make a mark on a horizontally-oriented, 10-point VAS labeled "no pain (zero point)" at the far left and "greatest pain (ten point)" at the far right.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Sup Yeom, MD. Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea